CLINICAL TRIAL: NCT04554836
Title: Modulation of the FOLFIRI-based Standard First-line Therapy With Cetuximab, Controlled by Monitoring the RAS (Rat Sarcoma) Mutation Load by Liquid Biopsy in RAS-mutated mCRC (Metastatic Colorectal Cancer): A Randomized Phase II Study With FOLFIRI-based First-line Therapy With or Without Intermittent Cetuximab (MoLiMoR)
Brief Title: MoLiMoR - A Study With FOLFIRI-based First-line Therapy With or Without Intermittent Cetuximab
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: TheraOp (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4213000
Record Dates: First submitted 2020-09-07; First posted 2020-09-18 (Actual); Results first posted 2025-06-08 (Actual); Last update posted 2025-06-08 (Actual); Status verified 2025-06

CONDITIONS: Adenocarcinoma of the Colon; Adenocarcinoma of the Rectum
Keywords: Left sided Adenocarcinoma of the Colon; RAS mutated
MeSH Terms: conditions — Colonic Neoplasms; Rectal Neoplasms | interventions — Cetuximab; IFL protocol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FOLFIRI + cetuximab (Experimental): Patients in Arm A will receive FOLFIRI + cetuximab until progressive disease (PD), unacceptable toxicity, withdrawal of informed consent or death, whatever occurs first. The recurrence of RAS-mutation without PD to switch back to FOLFIRI. In case of repeated conversion to RAS wild-type without PD, treatment will shift to FOLFIRI + cetuximab again, and so on. Switches of treatment will proceed until progressive disease (PD), unacceptable toxicity, withdrawal of informed consent or death, whatever occurs first.
  [FOLFIRI = Irinotecan, Folinic acid (racemic), Fluorouracil (5-FU)]
  Interventions: Drug: Cetuximab; Other: FOLFIRI
- FOLFIRI (Other): Patients in Arm B will continue therapy with FOLFIRI until PD, unacceptable toxicity, withdrawal of informed consent or death, whatever occurs first.
  Interventions: Other: FOLFIRI

INTERVENTIONS:
Drug: Cetuximab — Patients in Arm A will receive FOLFIRI +cetuximab.
  Arms: FOLFIRI + cetuximab
Other: FOLFIRI — Irinotecan, Folinic acid (racemic), Fluorouracil (5-FU)

SUMMARY:
This is an open-label, prospective, randomized, multicenter phase II trial that will evaluate the efficacy and safety of intermittent addition of cetuximab to a FOLFIRI-based first line therapy to patients with RAS (Rat sarcoma)-mutant mCRC (Metastatic colorectal cancer) diagnosis who convert to RAS wild-type using monitoring of the RAS mutation status by liquid biopsy.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed, UICC stage IV adenocarcinoma of the left-sided colon or rectum with metastases (metastatic colorectal cancer), primarily non-resectable, confirmed RAS mutations proven in the primary tumor or metastasis (KRAS ans NRAS exon 2, 3, 4)
* Age ≥ 18 years on day of signing informed consent
* No previous chemotherapy for metastatic disease (1- 2 cycles FOLFIRI or mFOLFIRI are permitted before enrolment until RAS status is determined)
* Patients suitable for chemotherapy administration
* ECOG (Eastern Cooperative Oncology Group) status 0-1
* Consent to liquid biopsy and mutation analysis
* Estimated life expectancy > 3 months
* Presence of at least one measurable reference lesion according to the RECIST 1.1 criteria (chest CT and abdominal CT 4 weeks or less before enrollment)
* Adequate bone marrow function defined as: Leukocytes 3.0 x 10 9/L with neutrophils 1.5 x 10 9/L, Thrombocytes 100 x 10 9/L, Hemoglobin 9 g/dL
* Adequate hepatic function defined as: Serum bilirubin 1.5 x ULN (Upper limit of normal), ALAT (Alanine-aminotransferase (= SGPT = serum glutamate pyruvate transaminase) and ASAT (aspartate-aminotransferase (= SGOT = serum glutamate oxalacetate transaminase) 2.5 x ULN (Upper limit of normal) (in the presence of hepatic metastases, ALAT and ASAT 5 x ULN)
* Adequate renal function: Creatinine clearance ≥ 50 mL/min
* Adequate cardiac function defined as Normal ECG and echocardiogram with a left ventricular ejection fraction (LVEF) of 55%
* INR (International normalized ratio) < 1.5 and aPTT (activated Partial thromboplastin time) < 1.5 x ULN (patients without anticoagulation). Therapeutic anticoagulation is allowed if INR and aPTT have remained stable within the therapeutic range for at least 2 weeks.
* Time interval of at least 6 months since last administration of any previous neoadjuvant/adjuvant chemotherapy or radiochemotherapy of the primary tumor in curative treatment intention to start of 1st line treatment
* Any relevant toxicities of prior treatments must have resolved to grade ≤ 1 according to the CTCAE (version 5), except alopecia
* Women of childbearing potential (WOCBP) should have a negative urine pregnancy test within 72 hours prior to receiving the first dose of study medication.
* Highly effective contraception for both male and female patients throughout the study and for at least 3 months after last dose of study medication administration if the risk of conception exists. Highly effective contraception has to be in line with the definition of the CTFG (Clinical Trial Facilitation Group) recommendation
* Signed written informed consent and capacity of understanding the informed consent

Exclusion Criteria:

* Right sided mCRC
* Primarily resectable metastases
* Previous chemotherapy for the colorectal cancer with the exception of adjuvant treatment, completed at least 6 months before entering the study (1- 2 cycles FOLFIRI or mFOLFIRI are permitted before enrolment)
* Patients with known brain metastases
* Symptomatic peritoneal carcinosis
* Progressive disease before randomization
* History of acute or subacute intestinal occlusion, inflammatory bowel disease, immune colitis or chronic diarrhea
* Grade II heart failure (NYHA classification), Myocardial infarction, balloon angioplasty (PTCA) with or without stenting, and cerebral vascular accident/stroke within the past 12 months before enrollment, unstable angina pectoris, serious cardiac arrhythmia according to investigator's judgment requiring medication
* Active infection with hepatitis B or C
* Medical or psychological impairments associated with restricted ability to give consent or not allowing conduct of the study
* Additional cancer; Exceptions include adequately treated basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or in situ cervical cancer that has undergone potentially curative therapy without evidence of recurrence
* Uncontrolled hypertension
* Marked proteinuria (nephrotic syndrome)
* Arterial thromboembolism or severe hemorrhage within 6 months prior to randomization (with the exception of tumor bleeding before tumor resection surgery)
* Hemorrhagic diathesis or tendency towards thrombosis
* Participation in a clinical study or experimental drug treatment within 30 days prior to study
* Known hypersensitivity or allergic reaction to any of the study medications
* Severe, non-healing wounds, ulcers, bone fractures or an infection requiring systemic therapy
* Known history of alcohol or drug abuse
* Complete dihydropyrimidine dehydrogenase (DPD) deficiency (phenotype and/or genotype test) (Patients with partial DPD deficiency may be included in this clinical trial at the discretion of the investigator and should receive a reduced starting 5-FU dose)
* Known glucuronidation deficiency (Gilbert's syndrome) (specific screening not required)
* Absent or restricted legal capacity
* For female patients only: Pregnancy (absence to be confirmed by ß-HCG test) or lactating

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2020-12-29 (Actual); Primary Completion 2024-06-11 (Actual); Study Completion 2024-06-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (4):
- Germany (4):
  - Universitätsklinikum Knappschaftskrankenhaus, Bochum
  - Onkologisches Zentrum (Dachau II), Dachau
  - Kliniken-Essen-Mitte Evang. Huyssens-Stiftung, Essen
  - Evangelisches Krankenhaus Hamm, Hamm

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Klein-Scory S, Wahner I, Maslova M, Al-Sewaidi Y, Pohl M, Mika T, Ladigan S, Schroers R, Baraniskin A. Evolution of RAS Mutational Status in Liquid Biopsies During First-Line Chemotherapy for Metastatic Colorectal Cancer. Front Oncol. 2020 Jul 16;10:1115. doi: 10.3389/fonc.2020.01115. eCollection 2020. PMID 32766143
- See also: Evolution of RAS Mutational Status in Liquid Biopsies During First-Line Chemotherapy for Metastatic Colorectal Cancer. — https://www.frontiersin.org/articles/10.3389/fonc.2020.01115/full?report=reader

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between September 2020 and July 2021 20 sites in Germany and 1 site in Austria screened patients. Of these, 4 sites randomized patients.
  1. Onkologisches Zentrum Donauwörth, Onkologisches Zentrum, Dachau
  2. Kliniken Essen-Mitte Evang. Huyssens-Stiftung, Klinik für internistische Onkologie/Hämatologie, Essen
  3. Universitätsklinikum Knappschaftskrankenhaus Bochum, Medizinische Klinik - Innere Medizin, Bochum
  4. Evangelisches Krankenhaus Hamm, Innere Medizin II, Hamm
Groups:
- FOLFIRI + Cetuximab: Patients in Arm A will receive FOLFIRI + cetuximab until progressive disease (PD), unacceptable toxicity, withdrawal of informed consent or death, whatever occurs first. The recurrence of RAS-mutation without PD to switch back to FOLFIRI. In case of repeated conversion to RAS wild-type without PD, treatment will shift to FOLFIRI + cetuximab again, and so on. Switches of treatment will proceed until progressive disease (PD), unacceptable toxicity, withdrawal of informed consent or death, whatever occurs first.
  [FOLFIRI = Irinotecan, Folinic acid (racemic), Fluorouracil (5-FU)]
  Cetuximab: Patients in Arm A will receive FOLFIRI +cetuximab.
  FOLFIRI: Irinotecan, Folinic acid (racemic), Fluorouracil (5-FU)
Period: Overall Study
Arm/Group | FOLFIRI + Cetuximab | FOLFIRI
Started | 4 | 2
Completed | 4 | 2
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: 129 patients were screened, 6 patients were randomized.
Groups:
- Total: Total of all reporting groups
Arm/Group | FOLFIRI + Cetuximab | FOLFIRI | Total
Number analyzed (Participants) | 4 | 2 | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 2 | 3
  >=65 years | 3 | 0 | 3
Age, Continuous [Mean (Full Range); unit: years] | 68.5 [62 to 80] | 46 [41 to 51] | 61 [41 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1
  Male | 3 | 2 | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 4 | 2 | 6
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Germany | 4 | 2 | 6

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS)
Description: Evaluation of efficacy in terms of progression free survival (PFS)
Time Frame: From date of randomization up to 24 months
Measure: Count of Participants; unit: Participants
Arm/Group | FOLFIRI + Cetuximab | FOLFIRI
Number analyzed (Participants) | 4 | 2
Participants | 0 | 0

2. Secondary Outcome: Overall Survival (OS)
Description: In experimental and control arms
Time Frame: From date of randomization up to 24 months.
Reporting Status: Not Posted

3. Secondary Outcome: Time to Failure of Treatment Strategy (TFTS)
Description: In experimental and control arms
Time Frame: After randomization up to 24 months.
Reporting Status: Not Posted

4. Secondary Outcome: PFS (Progression Free Survival) Rate
Description: In experimental and control arms
Time Frame: 1 year after date of randomization
Reporting Status: Not Posted

5. Secondary Outcome: Depth of Response
Description: In terms of reduction of tumor mass in experimental and control arms
Time Frame: From the start of the first line treatment in the study up to 24 months.
Reporting Status: Not Posted

6. Secondary Outcome: Metastasis Resections.
Description: In experimental and control arms.
Time Frame: From the start of the first line treatment in the study up to 24 months.
Reporting Status: Not Posted

7. Secondary Outcome: Objective Response Rate (ORR)
Description: Defined as patients with partial or complete response (CR or PR) in experimental and control arms
Time Frame: From the start of the first line treatment in the study up to 24 months.
Reporting Status: Not Posted

8. Secondary Outcome: Safety Profile
Description: According to CTCAE (Common Terminology Criteria of Adverse Events), Version 5.0 criteria in experimental and control arms.
Time Frame: From the date of signature of Informed Consent to 24 months.
Reporting Status: Not Posted

9. Secondary Outcome: Identification of Driver Mutations.
Description: In patients with progressive disease (PD) under cetuximab therapy who remain RAS (Rat sarcoma) wild-type in liquid biopsy.
Time Frame: From the start of the first line treatment in the study up to 24 months.
Reporting Status: Not Posted

10. Secondary Outcome: Comparison the Efficacy in Terms of Progression Free Survival (PFS)
Description: In patients with conversion to RAS (RAt sarcoma) wild-type in both ddPCR (Droplet Digital PCR) BEAMing with those patients showing conversion to RAS wild-type in ddPCR but not in BEAMing.
Time Frame: From the start of the first line treatment in the study up to 24 months.
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: up to 37 months (Consent of FPI until 30 days after last dose of study treatment)
Description: Adverse events have to be reported after informed consent until 30 days after last dose of study treatment. Then only adverse events which are causally related to study treatment have to be reported
Arm/Group | FOLFIRI + Cetuximab | FOLFIRI
All-Cause Mortality (participants affected / at risk) | 3/4 | 2/2
Serious Adverse Events (participants affected / at risk) | 3/4 | 0/2
Other Adverse Events (participants affected / at risk) | 4/4 | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FOLFIRI + Cetuximab (N=4) | FOLFIRI (N=2)
Colorectal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Hepatobiliary procedural complication (Hepatobiliary disorders) | 1 (1) | 0 (0)
Ileus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FOLFIRI + Cetuximab (N=4) | FOLFIRI (N=2)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Arrhythmia (Cardiac disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (2) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 2 (3) | 2 (3)
Dyschezia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Enteritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 3 (4) | 2 (3)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (2)
Fatigue (General disorders) | 1 (1) | 2 (2)
Pyrexia (General disorders) | 1 (1) | 1 (1)
Hypersensitivity (Immune system disorders) | 1 (1) | 0 (0)
Anorectal infection (Infections and infestations) | 0 (0) | 1 (1)
Infection (Infections and infestations) | 1 (1) | 0 (0)
Nail infection (Infections and infestations) | 1 (1) | 0 (0)
Skin infection (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Skin laceration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 1 (2)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1)
Blood bilirubin increased (Investigations) | 0 (0) | 1 (1)
Blood pressure abnormal (Investigations) | 1 (2) | 0 (0)
C-reactive protein increased (Investigations) | 2 (2) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (3)
Anticholinergic syndrome (Nervous system disorders) | 0 (0) | 1 (1)
Dysgeusia (Nervous system disorders) | 0 (0) | 1 (1)
Parosmia (Nervous system disorders) | 0 (0) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 1 (1)
Nightmare (Psychiatric disorders) | 1 (1) | 0 (0)
Stress (Psychiatric disorders) | 0 (0) | 1 (1)
Renal failure (Renal and urinary disorders) | 1 (1) | 0 (0)
Pelvic pain (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2)
Embolism (Vascular disorders) | 1 (1) | 0 (0)
Overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Therapy change (Surgical and medical procedures) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2021-03-09): https://cdn.clinicaltrials.gov/large-docs/36/NCT04554836/Prot_000.pdf
  • Statistical Analysis Plan (2024-09-13): https://cdn.clinicaltrials.gov/large-docs/36/NCT04554836/SAP_001.pdf